CLINICAL TRIAL: NCT01972698
Title: Focused Cardiac and Lung Ultrasound in Anesthesia/Critical Care - The Role of Self-directed Simulation-assisted Training Compared to a Traditional Supervised Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CCUS-Toronto01
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Education, Medical; Critical Care Ultrasonography
Keywords: Focused Cardiac Ultrasound; Lung Ultrasound; Simulation; Education; Web-based learning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-directed and simulation-assisted training (Experimental)
  Interventions: Other: Self-directed and simulation-assisted training
- Traditional apprenticeship training (Active Comparator)
  Interventions: Other: Traditional apprenticeship training

INTERVENTIONS:
Other: Self-directed and simulation-assisted training — All participants will attend an ultrasound introductory course (lectures and illustrative interactive cases).
  Participants randomized to the intervention group will undergo a completely self-directed lung and focused cardiac ultrasound curriculum.
  * A set of video-lectures on how to perform US on a critically ill patient (video-tutorials on image acquisition, troubleshooting, and pitfalls) will be provided.
  * Participant will have access to an ultrasound simulator.
  * Finally, participants in the intervention group will be asked to perform self-directed lung and focused cardiac ultrasound examinations on critically ill patients.
  An investigator will supervise the sessions but will not interfere with the self-learning process.
  - To support their learning, trainees will have access to on-line virtual FCU and LUS modules created by the Toronto General Hospital Department of Anesthesia Perioperative Interactive Education (http://pie.med.utoronto.ca/TTE/index.htm).
  Arms: Self-directed and simulation-assisted training
Other: Traditional apprenticeship training — All participants will attend an half-day ultrasound introductory course.
  * Participants randomized to the conventional group will initially attend 2-hour hands-on session on healthy volunteers, fully supervised by an expert critical care ultrasonographer (acquisition of basic knowledge with US machine settings and probe positioning and orientation, normal view acquisition, and identification of normal anatomical structures and landmarks).
  * Subsequently, participants will attend a 3-hours hands-on session on critically ill patients, fully supervised by an expert critical care ultrasonographer.
  Arms: Traditional apprenticeship training

SUMMARY:
The purpose of this study is to determine whether a self-directed and simulation-based lung ultrasound (LUS) and focused cardiac ultrasound (FCU) curriculum is efficacious on anesthesia trainees' image acquisition skills and diagnostic acumen. The investigators hypothesize that a self-directed and ultrasound-assisted LUS and FCU curriculum that includes video lectures, online teaching modules, an ultrasound simulator, and self-directed hands-on sessions on critically ill mechanically ventilated patients is effective in training novice ultrasonographers to obtain good quality images, to correctly interpret them, and to support clinical decision-making in critically ill patients.

Trainees will be randomized to fully supervised FCU hands-on sessions on healthy models and critically ill mechanically ventilated patients (control group - traditional apprenticeship model) or to a completely self-directed and simulation-based approach (intervention group).

To assess if this new self-directed and simulation-based ultrasound curriculum leads to adequate acquisition of competences (adequate image acquisition and interpretation) in novice ultrasonographers, trainees will have to perform a focused lung and cardiac assessment on a critically ill mechanically ventilated patient.

ELIGIBILITY:
Inclusion Criteria:

* PGY1 and PGY2 anesthesia resident at the University of Toronto

Exclusion Criteria:

* Previous training in lung ultrasound or FCU

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Difference between pre- and post-intervention image acquisition and interpretation skill (as compared to the benchmark exam). | ~4-5 months post-study enrolment, after completion of ultrasound training
  The quality of the images will be scored from 1 (worst) to 5 (best). The score will be based on the assessment of the quality of the image as well as an assessment of relevant cardiac structures included in each view.
  Difference between pre- and post-intervention image acquisition skills and knowledge as measured by:
  * Scanning time (total and per view)
  * Anatomy recognition
  * Items completion (%)
  * Image interpretation (Y/N for lung sliding, interstitial syndrome, pleural effusion, consolidation, pericardial fluid, LV global function, RV global function, intravascular volume assessment; total and per objective accuracy)
  * MCQs results (%) (Indication & Image interpretation assessment)
  * Video-interpretation of cases results (%) (Image interpretation & Clinical decision-making assessment)
  * Qualitative and quantitative analysis of survey results (dichotomic questions; graded criteria; e.g.10-point Likert scale)

SECONDARY OUTCOMES:
Differences between self-directed and simulation-assisted training and traditional apprenticeship training | ~4-5 months post-study enrolment, after completion of ultrasound training
  Difference between groups in image acquisition skills and knowledge as measured by:
  * Quality of images obtained (total and per view score)
  * Scanning time (total and per view)
  * Anatomy recognition (at least 4 structures identified/views for FCU, and 3 structures identified/LUS findings for LUS; max score 20 + 6)
  * Items completion (%)
  * Image interpretation (Y/N for lung sliding, interstitial syndrome, pleural effusion, consolidation, pericardial fluid, LV global function, RV global function, intravascular volume assessment; total and per objective accuracy)
  * MCQs results (%) (Indication & Image interpretation assessment)
  * Video-interpretation of cases results (%) (Image interpretation & Clinical decision-making assessment)
  * Qualitative and quantitative analysis of survey results (dichotomic questions; graded criteria; e.g.10-point Likert scale)

OTHER OUTCOMES:
Assessment of baseline visuo-spatial skill | ~4-5 months post-study enrolment, after completion of ultrasound training
  Visuo-spatial skill test scores compared to FCU outcomes related to technical proficiency gained (quality of images acquired; percent correct views obtained; scanning time; anatomy recognition).
Knowledge and skills retention at 3 months | ~4-5 months post-study enrolment, after completion of ultrasound training
  Difference between groups in image acquisition skill and knowledge as measured by:
  * Quality of images obtained (total and per view score)
  * Scanning time (total and per view)
  * Anatomy recognition (at least 4 structures identified/views for FCU, and 3 structures identified/LUS findings for LUS; max score 20 + 6)
  * Items completion (%)
  * Image interpretation (Y/N for lung sliding, interstitial syndrome, pleural effusion, consolidation, pericardial fluid, LV global function, RV global function, intravascular volume assessment; total and per objective accuracy)
  * MCQs results (%) (Indication & Image interpretation assessment)
  * Video-interpretation of cases results (%) (Image interpretation & Clinical decision-making assessment)
  * Qualitative and quantitative analysis of survey results (dichotomic questions; graded criteria; e.g.10-point Likert scale)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Abrahamson, MD, Principal Investigator — Unity Health Toronto; Han Kim, MD, Principal Investigator — Unity Health Toronto; Alberto Goffi, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Royse CF, Canty DJ, Faris J, Haji DL, Veltman M, Royse A. Core review: physician-performed ultrasound: the time has come for routine use in acute care medicine. Anesth Analg. 2012 Nov;115(5):1007-28. doi: 10.1213/ANE.0b013e31826a79c1. Epub 2012 Sep 25. PMID 23011559
- [Background] Labovitz AJ, Noble VE, Bierig M, Goldstein SA, Jones R, Kort S, Porter TR, Spencer KT, Tayal VS, Wei K. Focused cardiac ultrasound in the emergent setting: a consensus statement of the American Society of Echocardiography and American College of Emergency Physicians. J Am Soc Echocardiogr. 2010 Dec;23(12):1225-30. doi: 10.1016/j.echo.2010.10.005. PMID 21111923
- [Background] Spencer KT, Kimura BJ, Korcarz CE, Pellikka PA, Rahko PS, Siegel RJ. Focused cardiac ultrasound: recommendations from the American Society of Echocardiography. J Am Soc Echocardiogr. 2013 Jun;26(6):567-81. doi: 10.1016/j.echo.2013.04.001. No abstract available. PMID 23711341
- [Background] Expert Round Table on Ultrasound in ICU. International expert statement on training standards for critical care ultrasonography. Intensive Care Med. 2011 Jul;37(7):1077-83. doi: 10.1007/s00134-011-2246-9. Epub 2011 May 26. PMID 21614639
- [Background] Mayo PH, Beaulieu Y, Doelken P, Feller-Kopman D, Harrod C, Kaplan A, Oropello J, Vieillard-Baron A, Axler O, Lichtenstein D, Maury E, Slama M, Vignon P. American College of Chest Physicians/La Societe de Reanimation de Langue Francaise statement on competence in critical care ultrasonography. Chest. 2009 Apr;135(4):1050-1060. doi: 10.1378/chest.08-2305. Epub 2009 Feb 2. PMID 19188546
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Schmidt GA. ICU ultrasound. The coming boom. Chest. 2009 Jun;135(6):1407-1408. doi: 10.1378/chest.09-0502. No abstract available. PMID 19497889
- [Background] Neelankavil J, Howard-Quijano K, Hsieh TC, Ramsingh D, Scovotti JC, Chua JH, Ho JK, Mahajan A. Transthoracic echocardiography simulation is an efficient method to train anesthesiologists in basic transthoracic echocardiography skills. Anesth Analg. 2012 Nov;115(5):1042-51. doi: 10.1213/ANE.0b013e318265408f. Epub 2012 Jul 19. PMID 22822190